CLINICAL TRIAL: NCT02237443
Title: Ventilation by Mask Before and After the Administration of Neuromuscular Blockade: a Non-inferiority Trial
Brief Title: Mask Ventilation Before and After Neuromuscular Blockade
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Aaron Joffe, Assistant Professor, Anesthesiology & Pain Medicine, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 40262-D
Record Dates: First submitted 2014-08-28; First posted 2014-09-11 (Estimated); Last update posted 2015-04-09 (Estimated); Status verified 2015-04

CONDITIONS: Anesthesia
Keywords: Patient Safety
MeSH Terms: interventions — Rocuronium; Vecuronium Bromide; Succinylcholine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Post-induction (Other): Anesthesia is induced with propofol and mask ventilation is commenced after patient is unresponsive to a jaw thrust prior to administration of rocuronium, vecuronium bromide, or succinylcholine
  Interventions: Drug: Rocuronium; Drug: Vecuronium Bromide; Drug: Succinylcholine

INTERVENTIONS:
Drug: Rocuronium — Administration of a NMBD
Drug: Vecuronium Bromide — Administration of a NMBD
  Other Names: Vecuronium
Drug: Succinylcholine — Administration of a NMBD
  Other Names: Sux

SUMMARY:
Anesthesia providers are taught to "test" that they can properly ventilate a patient's lungs before administering a neuromuscular blocking drug (NMBD), rendering the patient apneic. This is a traditional teaching, not based on empirical evidence. The investigators primary hypothesis is that ventilation after the administration of NMBDs is non-inferior with that before their administration with respect to the composite safety endpoint of inadequate (MVi) and dead-space only (Vds) ventilation.

DETAILED DESCRIPTION:
The following will be carried out per routine standard of care:

The patient will be met in the pre-operative area by the attending anesthesiologist who interviews and examines the patient. A full explanation of the general anesthetic including risks and benefit will be given. Patients will be premedicated with 1-2 mg of midazolam at the discretion of the attending anesthesiologist. Once in the OR, standard American Society of Anesthesiology (ASA) monitors are established. At a minimum, this includes non-invasive monitoring of blood pressure by automated cuff, oxygen saturation via pulse oximetry, heart rate and rhythm by 3-lead continuous electrocardiographic tracing, core body temperature, expired carbon dioxide concentration, and depth of neuromuscular blockade when paralytic medications are used. Additional monitoring may be applied as deemed appropriate by the attending anesthesiologist on a case-by-case basis. At this time, the patient is given fentanyl 1-2 mcg/kg. After a period of breathing 100% oxygen by facemask (typically for 3 minutes or until the anesthesia monitor shows the exhaled concentration of oxygen to be >80%) and when the primary anesthesia team judges denitrogenation to be sufficient, anesthesia will be induced intravenously with propofol 2-3 mg/kg. Once the patient is unresponsive to a jaw thrust, the patient is ventilated via a facemask. If the anesthesia provider feels that ability to move air in and out of the patients lungs is difficult, the may reposition the mask on the patient's face, reposition the head, neck, or shoulders of the patient, or place a plastic oropharyngeal airway to maintain the mouth in an open position and to help keep the base of the tongue from obstructing the upper airway. A drug that causes muscle paralysis is given, which takes 1-5 minutes to work depending on the drug administered; during this period the patient continues to be ventilated by facemask. However, there is not standard for the timing of administration of the paralytic drugs as some anesthesia providers administer them near simultaneous to the administration of the other drugs used to induce anesthesia. Often, during this time, an inhaled anesthetic agent is started to avoid any gaps in the effect of the intravenous medications. Once the muscle relaxant works, a breathing tube is placed in the patient's windpipe, and ventilation occurs via the tube connected to a breathing machine.

The study deviates from the standard anesthesia care described above in the following ways:

Before the patient arrives in the operating room, a small plastic device called a pneumotachograph will be placed in-line between the facemask and the breathing circuit of the anesthesia machine. This allows measurements of airway pressure and volumes to be recorded in an accurate manner and later sent electronically to a computer for analysis. The in-line portion of the device is no larger than a typical circuit connector already used and does not hinder the performance of the anesthesia provider in any way. After routine intravenous induction, once the patient is unresponsive to a jaw thrust patients will be ventilated by facemask for 60 seconds. Breaths will be delivered using the breathing bag of the anesthesia circuit as would otherwise be performed. The airway managers will be asked to follow a treatment algorithm to resolve any difficulty encountered in providing mask ventilation. This algorithm represents common practice. After the initial 60 seconds, the medication to induce muscle paralysis will be given. A nerve stimulator placed on the patients wrist will then be turned on and will indicate when the medication has taken full effect and the patient is paralyzed. During this period of time, approximately 60-90 seconds, with the patients unconscious and apneic, their breathing will be supported as would otherwise be done. Post-paralysis, data collection will again begin and the anesthesia provider will start again breathing for the patient via a facemask as described in figure 2 for another 60 seconds. The operator will be blinded to the display on the ventilator machine, which provides information about the amount of air going in and out of the patients lungs, but will be able to monitor the patient's pertinent vital signs on the anesthesia machine. At all times, one member of the primary anesthesia team will have full access to all monitoring as would normally take place. After this time, the tracheal tube will be placed for the surgery.

Appropriate sizing of the adult facemask and oropharyngeal airway will be determined by the primary anesthesia team. All breaths will be delivered by hand ventilation using the breathing bag of the anesthesia machine. The returned tidal volume will be recorded for each minute of the study period from the pneumotachograph placed inline with the anesthesia circuit at the level of the mask/elbow connector interface as described above. The total time from induction to placement of a breathing tube will be 4-5 minutes and represents an additional minute of "study" time to the standard care. This timing was chosen as the investigators feel that it will provide sufficient information about ventilation volumes without unduly prolonging the anesthetic.

The study coordinator will remain in the room for the actual intubation to record its ease or difficulty per the report of the primary anesthesia provider. The act of placing the breathing tube is not part of the study protocol, however.

Data points to be collected:

Data regarding tidal volume, minute ventilation, airway pressures, and end-tidal carbon dioxide will be recorded directly by the in-line pneumotachograph and then loaded into an excel spreadsheet. No manual data collection will be necessary.

Data and Safety Monitoring Plan

The study may be terminated by the primary anesthesia team if the one or more of the following criteria are met:

1. Inadequate ventilation by clinical criteria (inadequate chest rise, no fogging in the mask, no positive tracing of end-tidal carbon dioxide and/or lack of measurable returned tidal volumes on).
2. Low oxygen saturation (< 90%).
3. If for any reason, the primary anesthesia team feel that in their clinical judgment, immediate tracheal intubation is warranted.

All unanticipated problems and adverse event will be recorded in the study sheet by a study coordinator. At the earliest time, each unanticipated problem and adverse event will be examined by at least 2 study investigators. In the event of an unanticipated problem of adverse effect (eg inadequate mask ventilation), back-up will be provided by the primary anesthesia team caring for the patient and may include placing a laryngeal mask airway or a surgical airway. These are the same provisions that would be made for any non-study case as mask ventilation by using one or two hands represents standard practice.

Statistical Considerations:

The investigators are aiming to show that administration of a neuromuscular blocking agent is "safe" with respect to mask ventilation. In other words, that the average exhaled tidal volume per breath over one minute after the administration of a NMBD will be non-inferior to that measured before their administration. At the time of the planning of this study, no studies had reported a mean±SD for tidal volumes before and after NMBDs. However, based upon a prior comparative trial of two different mask-hold techniques, the standard deviation (SD) of the average exhaled tidal volume after induction of anesthesia, using the anesthesia ventilator and a two-hand jaw-thrust mask hold technique was 130 mL. With the equivalence limit, d, set as 50 mL per breath, with a significance level (α) of 2.5% and a power (1-β) of 95%, a total sample size of 208 patients per group (before and after NMBD for a total sample of 416 study periods) were required. In other words, if there is truly no difference between the mask ventilation before and after NMBD, then 208 patients, each as their own control, are required to be 95% sure that the limits of a 2-sided 95% confidence interval will exclude a difference in means of >50 mL.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are 18 years or greater
* Present for elective surgery and
* Require placement of a breathing tube for their surgery

Exclusion Criteria:

* Patients will not be eligible if they are pregnant
* Are a minor
* Are a prisoner
* Have impaired decision-making capacity
* Have symptomatic untreated reflux
* Prior esophagectomy or hiatal hernia
* Vomiting within 24 hours of surgery
* Known oral or facial pathology making a proper mask fit unlikely
* Any condition for which the primary anesthesia team deems a rapid-sequence intubation to be appropriate
* Prior allergy or contraindication to receiving rocuronium, vecuronium, or succinylcholine.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2014-08; Primary Completion 2014-11 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Average exhaled title volumes | 2 minutes
  The difference in average exhaled volumes per breath between study periods before and after neuromuscular blocker administration.

SECONDARY OUTCOMES:
Minute ventilation (VE) | 2 minutes
  The total amount of gas exhaled per minute (the sum of all exhaled Vt over the study period)
Warter's scale | 2 minutes
  Clinico-physiologic scale for assessment of the difficulty of mask ventilation
Han's scale | 2 minutes
  Clinical scale for assessment of the difficulty of mask ventilation
Composite of difficult/impossible mask ventilation | 2 minutes
  The composite of difficult mask ventilation (DMV)/impossible mask ventilation (IMV) by Warter's scale and a volume definition of < 4 ml/kg predicted body weight or < 150 mL in total per breath on average

CONTACTS AND LOCATIONS:
Overall Officials: Aaron M Joffe, DO, Principal Investigator — University of Washington Department of Anesthesiology and Pain Medicine
Locations (1):
- Harborview Medical Center, Seattle, Washington, United States

REFERENCES:
- [Derived] Joffe AM, Ramaiah R, Donahue E, Galgon RE, Thilen SR, Spiekerman CF, Bhananker SM. Ventilation by mask before and after the administration of neuromuscular blockade: a pragmatic non-inferiority trial. BMC Anesthesiol. 2015 Oct 6;15:134. doi: 10.1186/s12871-015-0111-z. PMID 26444853